CLINICAL TRIAL: NCT02487264
Title: Analysis of the Status, Treatment and Outcomes of Rib Fractures
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Julia Caldwell, Assistant Professor of Anesthesiology and Pain Medicine, Milton S. Hershey Medical Center
Other Study IDs: 1125
Record Dates: First submitted 2015-04-05; First posted 2015-07-01 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Rib Fracture; Trauma
MeSH Terms: conditions — Rib Fractures; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A retrospective analysis of all patient presenting with multiple rib fractures to the emergency room of Penn State Hershey Medical Center between 2010-2012. Patient demographics, cause of fracture, outcomes, chronic medical conditions, vital signs, length of stay, pain levels and treatment, and sequelae will be recorded and analyzed.

DETAILED DESCRIPTION:
This is a retrospective chart review with follow-up phone calls.

The initial part of the study will be a retrospective chart review. For this chart review study, the following data elements will be entered for each participant.

The investigators will perform a retrospective study of patients who have been treated for rib fractures at Penn State Hershey Medical Center (PSHMC). The time period of review will be 1/10/10 - 1/10/12 until 1500 cases have been reviewed. Data collected will be:

* Patient Medical Record Number (MRN)
* Name
* Phone number
* length of stay (admit and discharge date)
* Number of rib fractures per patient
* Cause of rib fracture
* Characteristics of the fracture (unilateral versus bilateral and multiple versus single)
* Pain management used for the rib fracture including pain interventions, medications and all pain scores
* Complications attributable to the rib fracture, including:

  1. Shortness of Breath (SOB)
  2. Hemothorax,
  3. Pneumothorax
  4. Flail chest
  5. Intubation required
  6. Mechanical ventilation required
  7. Opioids required for pain
  8. Chest tube placement required
* Sequelae of rib fracture, including:

  1. Acute Respiratory Deficiency Syndrome (ARDS)
  2. Pneumonia
  3. Death
  4. chronic pain
  5. delayed subclavian vessel thrombosis
  6. aortic aneurysm
  7. tracheobronchial fistula
  8. thoracic outlet syndrome
  9. Horner's syndrome
* Clinical history of

  1. Rib fractures
  2. Other fractures
  3. Osteoporosis
  4. Chronic Obstructive Pulmonary Disease (COPD)
  5. Cancer
  6. Myocardial Infarction (MI) / Coronary Artery Disease (CAD)
  7. Arthritis
  8. Parkinson's disease
* Patient characteristics:

  1. Age
  2. Gender
  3. Race
  4. Body Mass Index (BMI)
  5. Alcohol use
  6. Smoking status
  7. Marital status
  8. Education
  9. Initial blood pressure

7.2.2 Follow-up phone calls

The investigators will then attempt to call the patients for follow-up information using a summary explanation of research phone script to obtain the following information:

1. pain score
2. quality of life via the EuroQol's quality of life survey :EQ-5D-3L questionnaire
3. pain meds

ELIGIBILITY:
Inclusion Criteria:

* must have above and be notated in our medical record

Exclusion Criteria:

* missing data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presenting during 2010-2012 with multiple rib fractures to PSHMC emergency department
Sampling Method: Non-Probability Sample
Enrollment: 921 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2017-12-14 (Actual)

PRIMARY OUTCOMES:
Types and treatment of Rib Fractures | Past 4 years
  * Characteristics of the fracture (unilateral versus bilateral and multiple versus single)
  * Pain management used for the rib fracture including pain interventions, medications and all pain scores

SECONDARY OUTCOMES:
sequelae and complications from rib fractures | Past 4 years
  sequelae and complications in patients presenting with rib fractures: •Complications attributable to the rib fracture, including:
  1. Shortness of Breath (SOB)
  2. Hemothorax,
  3. Pneumothorax
  4. Flail chest
  5. Intubation required
  6. Mechanical ventilation required
  7. Opioids required for pain
  8. Chest tube placement required
Pain levels | Past 4 years
Patient Characteristics | past 4 years
  * Clinical history of
    1. Rib fractures
    2. Other fractures
    3. Osteoporosis
    4. Chronic Obstructive Pulmonary Disease (COPD)
    5. Cancer
    6. Myocardial Infarction (MI) / Coronary Artery Disease (CAD)
    7. Arthritis
    8. Parkinson's disease
  * Patient characteristics:
    1. Age
    2. Gender
    3. Race
    4. Body Mass Index (BMI)
    5. Alcohol use
    6. Smoking status
    7. Marital status
    8. Education
    9. Initial blood pressure
Current patient quality of life as assessed by telephone survey | past 4 years
  Follow-up phone calls
  The investigators will then attempt to call the patients for follow-up information using a summary explanation of research phone script to obtain the following information:
  1. pain score
  2. quality of life via the EuroQol's quality of life survey :EQ-5D-3L questionnaire
  3. pain meds